CLINICAL TRIAL: NCT00483327
Title: Prospective Trial of Conservative Management of Atypical Endometrial Hyperplasia and Well to Moderately Differentiated Endometrial Carcinoma Using Megestrol Acetate
Brief Title: Management of Atypical Endometrial Hyperplasia and Endometrial Carcinoma Using Megestrol Acetate
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-685
Record Dates: First submitted 2007-06-05; First posted 2007-06-07 (Estimated); Results first posted 2016-07-01 (Estimated); Last update posted 2018-04-04 (Actual); Status verified 2018-03

CONDITIONS: Atypical Endometrial Hyperplasia; Endometrial Carcinoma
Keywords: Well; Moderately; Differentiated
MeSH Terms: conditions — Endometrial Hyperplasia; Endometrial Neoplasms | interventions — Megestrol Acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Megestrol Acetate (Experimental): 80 mg (2 tablets) orally at breakfast, 80 mg at dinner for at least 12 weeks and up to 2 years.
  Interventions: Drug: Megestrol Acetate

INTERVENTIONS:
Drug: Megestrol Acetate
  Other Names: Megace

SUMMARY:
The purpose of this trial is to study the efficacy, toxicity, and tolerability of a standard hormonal regimen of Megestrol Acetate (Megace) in the treatment of Atypical Endometrial Hyperplasia or well to moderately differentiated endometrial carcinoma.

DETAILED DESCRIPTION:
The trial's objectives are to study the efficacy, defined as complete pathologic resolution of disease, of a standard hormonal regimen with the progestin Megace for the treatment of atypical endometrial hyperplasia or well or moderately differentiated endometrial carcinoma in women desiring conservative medical management of these conditions in the Women's Cancer Program at the NYU School of Medicine and at the Bellevue Gynecologic Oncology clinics.

The major endpoint is pathologic complete response (pCR). For the purposes of this study, patients will be reevaluated for response every 12 weeks until complete response. Response will be assessed within 4 weeks of completion of 12 weeks of Megace, by endometrial biopsy or dilation and curettage (D&C)/hysteroscopy. An endometrial biopsy is sufficient to document progressive, stable disease or partial response. A D&C is necessary to confirm complete response.

Patients whose disease has completely responded will discontinue treatment and be encouraged to pursue fertility. Those not desiring immediate fertility will be placed on low dose oral contraceptive pills for at least 6 months. Patients who have had either a partial response or stable disease will be recounseled and offered continued medical management or surgical therapy. Patients whose disease has progressed will be offered definitive surgical management. Those patients declining surgery will still be followed on study.

ELIGIBILITY:
Inclusion Criteria:

* Women with a diagnosis of atypical endometrial hyperplasia or G1 or G2 endometrial carcinoma confirmed by an New York University (NYU) pathologist desiring medical management will be eligible. The diagnosis may be obtained either by endometrial biopsy or D&C. If diagnosis has been made outside of NYU, slides must be available for review.
* Age > = 18 years.
* Life expectancy of greater than 12 months.
* Gynecologic Oncology Group (GOG) performance status score of 0, 1 or 2
* Patients must have normal organ and marrow function as defined below:

  * leukocytes > = 3,000/mcL
  * platelets > = 100,000/mcL
  * total bilirubin within normal institutional limits
  * AST(SGOT)/ALT(SGPT) no greater than 2.5 X institutional upper limit of Normal
  * glucose < 200 mg/dl
  * creatinine within normal institutional limits OR
  * creatinine clearance > = 60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal
* Eligibility of patients receiving any medications or substances known to affect or with the potential to affect the activity or pharmacokinetics of Megace will be determined following review of their case by the Principal Investigator.
* The effects of Megace on the developing human fetus at the recommended therapeutic dose are unknown. For this reason and because Megace is known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients with a histological diagnosis of clear cell, papillary serous or poorly differentiated (G3) endometrial carcinoma.
* Patients with cancer have an MRI showing evidence of extrauterine spread or myometrial invasion.
* Presence of US findings suspicious for ovarian malignancy, unclear endometrial primary or recurrent endometrial cancer.
* Patients receiving other investigational agents.
* Patients with a history of a previous thrombotic event, known thrombophilic condition or poorly controlled diabetes.
* Patients with a history of breast cancer or other hormonally responsive malignancy.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because Megace has the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with Megace, breastfeeding should be discontinued if the mother is treated with Megace.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2007-06; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie V Blank, M.D., Principal Investigator — New York University
Locations (2):
- United States (2):
  - Bellevue Hospital, New York, New York
  - NYU Cancer Center, New York, New York

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From May 2007 to April 2012, total 31 patients were recruited to the study from New York University medical center and its affiliated hospitals.
Pre-assignment Details: One patient withdrew before the start of the treatment; ony 30 patients started the treatment.
Period: Overall Study
Arm/Group | Megestrol Acetate
Started | 30
Completed | 20
Not Completed | 10
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 3
Not completed — Lost to Follow-up | 4
Not completed — Patient Non Compliance | 2

BASELINE CHARACTERISTICS:
Population: All the patients enrolled to the study (including one who withdrew before the start of treatment)
Arm/Group | Megestrol Acetate
Number analyzed (Participants) | 31
Age, Customized [Number; unit: participants]
  18-24 years | 1
  25-34 years | 12
  35-44 years | 12
  45-54 years | 4
  55-64 yeras | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 6
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 18
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 31
Histological Diagnosis [Number; unit: participants]
  Atypical endometrial hyperplasia | 20
  FIGO Grade 1 endometrioid carcinoma | 9
  FIGO Grade 2 endometrioid carcinoma | 2

OUTCOME MEASURES:

1. Primary Outcome: Best Pathologic Responses
Description: Patients are evaluated every 12 weeks while on treatment. The response is evaluated by endometrial biopsy or dilation and curettage (D&C)/hysteroscopy. Complete response (CR) is defined as endometrial sampling is read as normal or proliferative endometrium. Partial response (PR) is defined as the biopsy sample has changed on the endometrial evaluation scale by at least one level towards normal. Stable disease (SD) is defined as no change in pathology between the index and follow-up sample. Progressive disease (PD) is defined the follow-up sample has changed towards neoplasia on the endometrial evaluation scale by at least one level or imaging is concerning for myometrial invasion or extrauterine disease such that conservative management is no longer medically appropriate.
Time Frame: up to 24 months
Population: Patient who were able to complete at least one full course (12 weeks) of treatment
Measure: Number; unit: participants
Arm/Group | Megestrol Acetate
Number analyzed (Participants) | 30
participants
  Pathologic CR | 17
  Unconfirmed CR | 4
  PR | 6
  SD | 1
  PD | 2

2. Secondary Outcome: Toxicity and Tolerability
Description: Patients with adverse events (AEs) which were possibly, probably, or definitely related to the treatment. AEs were evaluated according to Common Terminology Criteria for Adverse Events (CTCAE) 3.
Time Frame: up to 36 months
Population: Any patient with at least one dose of treatment.
Measure: Number; unit: participants
Groups:
- Grade 1 or 2; Grade 3: 80 mg (2 tablets) orally at breakfast, 80 mg at dinner for at least 12 weeks and up to 2 years.
Arm/Group | Grade 1 or 2 | Grade 3
Number analyzed (Participants) | 30 | 30
participants
  Weight gain | 9 | 0
  Mood alterations | 4 | 0
  Headache | 5 | 2
  Thromboembolic event | 0 | 1
  Carpal tunnel syndrome | 1 | 0
  Weakness | 1 | 0
  Vaginal Spotting | 6 | 0
  Vaginal Pain | 1 | 0
  Nausea | 6 | 0
  Insomnia | 4 | 0
  Fatigue | 6 | 0
  Abdominal Pain | 2 | 0
  Constipation | 3 | 0
  Increased Appetite | 4 | 0
  Depression | 3 | 0
  Bloating | 4 | 0

3. Secondary Outcome: Duration of Response
Description: For each patient, assessed every 12 weeks during treatment and every 6 months during follow-up.
Time Frame: up to 4 years
Population: The original PI for this study is no longer at our institution. Additionally, co-investigator has stated that this data was not collected and therefore not analyzed. This information is not available for reporting as it does not exist.
Arm/Group | Grade 1 or 2 | Grade 3
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Number of Women Who Became Pregnant
Time Frame: up to 3 years after the treatment for each patient
Population: Only 7 participants in the trial pursued pregnancy.
Measure: Number; unit: participants
Arm/Group | Megestrol Acetate
Number analyzed (Participants) | 7
participants | 3

ADVERSE EVENTS:
Description: All the adverse events are reported here regardless of attribution.
Arm/Group | Megestrol Acetate
Serious Adverse Events (participants affected / at risk) | 1/30
Other Adverse Events (participants affected / at risk) | 29/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Megestrol Acetate (N=30)
Thrombosis/thrombus/embolism (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Megestrol Acetate (N=30)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 1
Anorexia (Gastrointestinal disorders) | 1
Confusion (Nervous system disorders) | 1
Constipation (Gastrointestinal disorders) | 3
Constitutional Symptoms - Other: thirst (General disorders) | 3
Cystitis (Renal and urinary disorders) | 1
Dermatology/Skin - Other: skin peeling (Skin and subcutaneous tissue disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Distension/bloating, abdominal (Gastrointestinal disorders) | 5
Dizziness (Nervous system disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 2
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 1
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 4
Edema: head and neck: (Blood and lymphatic system disorders) | 1
Fatigue (asthenia, lethargy, malaise) (General disorders) | 7
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Flu-like syndrome (General disorders) | 1
Flushing (Skin and subcutaneous tissue disorders) | 1
Gastrointestinal - Other: Increased Appetite (Gastrointestinal disorders) | 4
Glucose, serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 1
Hemorrhage, GU: Vagina (Reproductive system and breast disorders) | 17
Hemorrhage/bleeding associated with surgery, intra-operative or postoperative (Injury, poisoning and procedural complications) | 1
Hot flashes/flushes (Endocrine disorders) | 3
Hypertension (Cardiac disorders) | 2
Hypotension (Cardiac disorders) | 1
Insomnia (General disorders) | 4
Irregular menses (change from baseline) (Reproductive system and breast disorders) | 1
Libido (Reproductive system and breast disorders) | 1
Memory impairment (Nervous system disorders) | 1
Mood alteration: Agitation (Nervous system disorders) | 1
Mood alteration: Anxiety (Nervous system disorders) | 3
Mood alteration: Depression (Nervous system disorders) | 5
Muscle weakness, generalized or specific area (not due to neuropathy): Whole body/generalized (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal/Soft Tissue - Other: Spasm (Musculoskeletal and connective tissue disorders) | 1
Nausea (Gastrointestinal disorders) | 7
Neuropathy: cranial: CN V Motor-jaw muscles; Sensory-facial (Nervous system disorders) | 1
Neuropathy: sensory (Nervous system disorders) | 3
Odor (patient odor) (General disorders) | 1
Pain - Other: side of body (General disorders) | 2
Pain: Abdomen NOS (Gastrointestinal disorders) | 7
Pain: Back (Musculoskeletal and connective tissue disorders) | 3
Pain: Chest/thorax NOS (Respiratory, thoracic and mediastinal disorders) | 2
Pain: Extremity-limb (Musculoskeletal and connective tissue disorders) | 1
Pain: Head/headache (Nervous system disorders) | 7
Pain: Muscle (Musculoskeletal and connective tissue disorders) | 1
Pain: Neuralgia/peripheral nerve (Nervous system disorders) | 1
Pain: Pelvis (Reproductive system and breast disorders) | 1
Pain: Pleura (Respiratory, thoracic and mediastinal disorders) | 1
Pain: Throat/pharynx/larynx (Respiratory, thoracic and mediastinal disorders) | 2
Pain: Vagina (Reproductive system and breast disorders) | 1
Proteinuria (Metabolism and nutrition disorders) | 1
Pruritus/itching (Skin and subcutaneous tissue disorders) | 1
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 1
Renal/Genitourinary - Other: Burning With Urination (Renal and urinary disorders) | 1
Rigors/chills (General disorders) | 1
Sweating (diaphoresis) (General disorders) | 2
Urinary frequency/urgency (Renal and urinary disorders) | 4
Urticaria (hives, welts, wheals) (Immune system disorders) | 1
Vaginal discharge (non-infectious) (Reproductive system and breast disorders) | 2
Vomiting (Gastrointestinal disorders) | 1
Weight gain (General disorders) | 9
Dermatology/Skin - Other: blister (Skin and subcutaneous tissue disorders) | 1
Pain: Pain NOS (General disorders) | 1
pain: stomach (Gastrointestinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes